CLINICAL TRIAL: NCT00160823
Title: Impact of a Self-Administered Information Leaflet on Adequacy of Colonic Cleansing for in-Hospital
Brief Title: Impact of a Self-Administered Information Leaflet on Adequacy of Colonic Cleansing for in-Hospital Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: 04-147
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Colonoscopy
Keywords: Colon cleansing; Quality; Cost-effectiveness

INTERVENTIONS:
Procedure: Self-administered leaflet

SUMMARY:
The quality of colon cleansing has a major impact on efficiency and cost of colonoscopy. A hand-out was made to instruct and motivate patients to adequately clean the bowel before colonoscopy.

The aim of the study is to compare adequacy of bowel cleansing in hospitalized patients receiving the hand-out or not on the day before colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Total colonoscopy scheduled during hospital stay in the Hôpital Universitaire de Genève (excluding dependencies);
* Informed consent for inclusion in the study signed by the patient;
* Ability to read and write at least one of the following languages : French, English, Spanish, Portuguese.

Exclusion Criteria:

* Colonoscopy scheduled under general anesthesia;
* Occupation inside the healthcare professions;
* Previous colonoscopy, colostomy or colectomy;
* Megacolon or idiopathic pseudo-obstruction.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2005-09

PRIMARY OUTCOMES:
Quality of overall colon cleansing

SECONDARY OUTCOMES:
Quality of cleansing in the ascending colon,
Frequency of inadequate preparation and of failed procedure,
Time to intubate the caecum,
Cost-effectiveness of the self-administered leaflet,
Patient compliance with the self-administered leaflet,
Patient comfort with the colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Dumonceau, MD,PhD, Study Chair — University Hospital, Geneva
Locations (1):
- Gastroenterology and Hepatology Division, University Hospital of Geneva, Geneva, Switzerland